CLINICAL TRIAL: NCT02548390
Title: A Phase 1/1b, Multicenter, Open-Label Study of Intravenous RXDX-107 in Adult Patients With Locally Advanced or Metastatic Solid Cancer
Brief Title: Study of Intravenous RXDX-107 in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXDX-107-01
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Solid Tumor
Keywords: Phase 1/1b; open-label; dose-escalation; pharmacokinetics; solid tumor; metastatic cancer; chemotherapy; nano formulation; alkylator
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RXDX-107 (Experimental)
  Interventions: Drug: RXDX-107

INTERVENTIONS:
Drug: RXDX-107 — Subjects in this study will receive RXDX-107 intravenously at dose levels specified for their respective dose cohorts. Dosing will begin at 25 mg/m2 on Day 1 and Day 2 of a 28-day cycle and will escalate until the maximum tolerated dose (MTD) or (RP2D) is determined. An additional schedule of administration of RXDX-107 on Day 1 of a 28 day cycle may be assessed. Cycles will be repeated in four-week (28 day) intervals for up to 6 cycles or until progression of disease, unacceptable toxicity, or another discontinuation criterion is met.

SUMMARY:
This is an open-label, Phase I/Ib, dose escalation study of intravenous RXDX-107 administered to subjects with advanced solid tumors. The study is designed to explore the safety, maximum tolerated dose (MTD), pharmacokinetics, pharmacodynamics, and preliminary clinical activity of RXDX-107 and to define a recommended Phase 2 dose (RP2D)

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed relapsed or refractory locally advanced or metastatic solid cancer for whom no standard therapy is considered appropriate, or for whom standard therapy is considered intolerable.
2. >18 years of age.
3. ECOG performance status of 0 or 1.
4. Life expectancy of at least 3 months.
5. Received the last dose of previous treatment / therapy before Day 1 of cycle 1:

   * 28 days for cytotoxic chemotherapy, immunotherapy, whole brain radiotherapy, anticonvulsive therapy, stereotactic radiosurgery and major surgery
   * 42 days for nitrosureas, mitomycin C, and liposomal anthracycline
   * 14 days for non-cytotoxic cancer therapies and radiotherapy
6. Recovered from all toxic effects (excluding alopecia) of any prior anti-cancer therapy to Grade ≤ 1 or to the baseline laboratory values.
7. Adequate organ function and baseline laboratory values
8. Women of childbearing potential must have a negative serum pregnancy

Phase 1b: Patient must have measurable disease

Exclusion Criteria:

1. Receiving other experimental therapy
2. Known symptomatic brain mets or leptomeningeal involvement
3. Myocardial infarction in the previous 12 weeks. Active ischemia or any other uncontrolled cardiac condition such as angina pectoris, significant cardiac arrhythmia requiring therapy, uncontrolled hypertension, or CHF.
4. Another concurrent illness which would preclude study conduct and assessment, uncontrolled: medical condition, active infection, risk of bleeding, diabetes mellitus, or pulmonary disease, or alcoholic liver disease, or primary biliary cirrhosis.
5. Malignancy within 3 years or active disease requiring treatment other than the target cancer. The exceptions are prostate cancer (Gleason grade < 6 with normalized PSA levels), treated in situ cervical, breast carcinoma, squamous or basal cell skin cancer.
6. Any condition that may compromise the ability to give written informed consent or to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Phase 1: Safety profile of RXDX-107 as characterized by Adverse Events, ECG and laboratory abnormalities | Approx. 1 year
  AEs, ECG and Labs assessed according to NCI CTCAE V4.0
Phase 1: Maximum observed plasma drug concentration (Cmax) | Approx. 1 year
  Plasma concentrations obtained following the dose on Day 1 (and from the dose on Day 2 in patients receiving the Day 1 and Day 2 schedule)
Phase 1: Time to Cmax, by inspection (tmax) | Approx. 1 year
  Plasma concentrations obtained following the dose on Day 1 (and from the dose on Day 2 in patients receiving the Day 1 and Day 2 schedule)
Phase 1: Area under the drug concentration by time curve (AUC) | Approx. 1 year
  From time 0 to the time of the last detectable plasma concentration (AUC0-t)
Phase 1: Apparent plasma terminal elimination rate constant (λz) and associated terminal half life (t½) | Approx. 1 year
  Plasma concentrations obtained following the dose on Day 1 (and from the dose on Day 2 in patients receiving the Day 1 and Day 2 schedule)
Phase 1: Plasma clearance (CL) | Approx. 1 year
  Plasma concentrations obtained following the dose on Day 1 (and from the dose on Day 2 in patients receiving the Day 1 and Day 2 schedule)
Phase 1: Volume of distribution (Vz) | Approx. 1 year
  Plasma concentrations obtained following the dose on Day 1 (and from the dose on Day 2 in patients receiving the Day 1 and Day 2 schedule)
Phase 1: Maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) | Approx. 6 months
Phase 1b: Confirm RP2D | Approx. 1 year
  Number of participants with Treatment-related AEs, Labs changes from baseline, and QTc interval changes from baseline assessed according to NCI CTCAE V4.0, concomitant medication usage, including all supportive care provided, and preliminary anti-tumor activity per RECIST v1.1 as assessed by Investigator

SECONDARY OUTCOMES:
Antitumor activity of RXDX-107 as measured by Objective Response Rate (ORR) | Approx. 1 year
  Per RECIST v1.1 as assessed by Investigator

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Florida Cancer Specialists, Sarasota, Florida
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - Tennessee Oncology, LLC, Nashville, Tennessee